CLINICAL TRIAL: NCT00839722
Title: Fertility After Uterine Artery Embolisation for the Treatment of Leiomyomas
Acronym: EFU
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P071006
Record Dates: First submitted 2009-02-06; First posted 2009-02-09 (Estimated); Last update posted 2019-06-20 (Actual); Status verified 2011-06

CONDITIONS: Leiomyomas; Fertility
Keywords: Uterine embolization; leiomyomas; fertility; myomectomies
MeSH Terms: conditions — Leiomyoma | interventions — Embolization, Therapeutic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): fertility after embolization
  Interventions: Procedure: embolization

INTERVENTIONS:
Procedure: embolization — fertility after embolization

SUMMARY:
The main goal of this study is to evaluate spontaneous fertility after uterine leiomyomas embolization, in women between 18 and 40 years old.

DETAILED DESCRIPTION:
Uterine artery embolization (UAE) is an effective treatment for leiomyomas, that has been proposed to replace hysterectomy in women who don't want any more pregnancy. Few authors have investigated the results of UAE in women desiring subsequent pregnancy. It might represents an alternative to multiples myomectomies by laparotomy , which results on postoperative fertility remain disappointing. The main goal of this study is to evaluate spontaneous fertility after uterine embolization, in women between 18 and 40 years old. The functional outcome, the efficiency, complications and side-effects of UAE will be also reported especially on the reproduction function. This will be an open prospective, multicentric, non-randomized, interventional study. Within the context of an experimental phase II essay, an optimal Simon plan with 2 stages is required. The current study is the first step. It will include 30 patients treated in the Gynecology departments of Pr MADELENAT and Pr Mathieu CAPUTO (BICHAT Hospital, Paris) and Pr Ville (Poissy Hospital, Poissy). Preliminary results will be reported at 1 year postoperative which correspond to the participation period of 15 months and the total follow-up period will be 2 years. Inclusion criteria will be the women whom multiples myomectomies by laparotomy would be necessary, with symptomatic myoma and an immediate wish of pregnancy. The number of first pregnancies among women who try to be pregnant (conception rate) and among all women (fertility rate) will be calculated. The effects of the embolisation on the genital physiology, the leiomyomas and the ovarian function will be evaluated by questionaries, clinical examination, biology exams (hormones), ultrasound and IRM at 3, 6 and 12 months, and coelioscopy and hysteroscopy at 3 months. The pregnancy progress will be evaluated in a longer study.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years and ≤ 40 years
* diffuse POLYMYOMATOSIS or recurrent POLYMYOMATOSIS after surgery requiring multiple myomectomies by laparotomies i.e. at least 3 fibroids of significant diameter (including 1 fibroid longer than 3 cm using ultrasound)
* symptomatic fibroids causing chronic pelvic pain and/or pelvic pressure and/or haemorrhage genital
* immediate desire for future pregnancy without indication for assisted medical reproduction (bilateral hydrosalpinx, male infertility)
* covered by french health insurance
* patient knowing to read and understanding French
* patient signing of an informed consent form, after appropriate information has been provided

Exclusion Criteria:

* evolutionary pregnancy
* medical emergency situation
* Contraindication by the surgery or Uterine Artery Embolisation : allergy, severe renal failure, immune system deficiency or anesthesic
* age > 40 years
* fibroids accessible to laparoscopies removal (less than 3 fibroids measuring 3 cm or 1 dominant fibroid measuring 8 cm) or hysteroscopies resection (submucous fibroids type 0 or I according to DONNEZ'S classification) or abdominal myomectomy indicated by large volume single intramural or subserosal fibroid
* abnormal hormonal profile at day 3 of the cycle evaluated during a pluridisciplinary consultation
* Male infertility requiring management for assisted medically reproduction (systematic
* spermograms will be obtained in routinely)
* amenorrhea
* visible hydrosalpinx for ultrasonography or MRI
* no explored an adnexal mass
* diffuse adenomyosis as the dominant disease
* no affiliation of social coverage
* bad comprehension of french preventing an informed consent form or information of self questionnaires
* social situation posing to difficulty of follow-up

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2009-02; Primary Completion 2011-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
The main goal of this study is to evaluate spontaneous fertility after uterine embolization, in women between 18 and 40 years old | 18 MONTHS

SECONDARY OUTCOMES:
The functional outcome, the efficiency, complications and side-effects of UAE will be also reported especially on the reproduction function | 18 MONTHS

CONTACTS AND LOCATIONS:
Overall Officials: Jean Pierre PELAGE, PUPH, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hopital Poissy St Germain En Laye, Poissy, France